CLINICAL TRIAL: NCT07084272
Title: A Comparison Study of ACD-A and EDTA Anticoagulation of Platelet-rich Plasma: Yields and Platelet Distribution
Brief Title: PRP Yield and Platelet Distribution With EDTA
Status: Not yet recruiting | Type: Observational
Sponsor: Harrison, Theodore, M.D. (Individual)
Responsible Party: Principal Investigator, Theodore Harrison, MD, MD, Harrison, Theodore, M.D.
Other Study IDs: PRPEDTA
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: PRP
Keywords: PRP; ACD-A; EDTA; platelets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will test and compare the platelet distribution after centrifugation and the platelet yield of ACD-A and EDTA anticoagulated blood

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* blood dyscrasias

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients receiving PRP treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet yield | 5 months
  fraction of platelets recovered in PRP
Platelet yield | 5 months
  percent of platelets in PRP compared to original blood sample

IPD SHARING:
Plan to Share IPD: No
too much administrative burden